CLINICAL TRIAL: NCT00412009
Title: Investigation of a Novel Approach to Improve Adherence to Treatment and Treatment Success Rates for Tuberculosis Patients in Senegal
Brief Title: Investigation of a Novel Approach to Improve Treatment Success Rates for Tuberculosis Patients in Senegal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAL+ 2671
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-12

CONDITIONS: Tuberculosis
Keywords: tuberculosis; control; treatment; adherence
MeSH Terms: conditions — Tuberculosis

INTERVENTIONS:
Procedure: Comprehensive package of activities

SUMMARY:
Tuberculosis (TB) patients who receive inadequate treatment or do not complete therapy are more likely to remain infectious, thus contributing to the continuous spread of TB infection in communities. Despite the widespread use of Directly Observed Therapy, defaulters remain an important problem in TB control programmes. In Sénégal, defaulters rate reach 30%, which is hampering dramatically the effectiveness of control. New strategies to deliver treatment to TB patients and ensure proper adherence that are adapted to the local situations are urgently needed.

Objectives

The overall objective of the project is to improve tuberculosis treatment success rates in Sénégal. The specific objectives are:

1. to assess the current situation of tuberculosis (TB) in Sénégal
2. to identify the determinants of cure,
3. to develop measures to improve patient's compliance with the treatment that are adapted to the local situation, acceptable, affordable and sustainable
4. to evaluate the impact of these measures on TB control.

Methods

The proposed research seeks to develop and test innovative methods to improve cure rates in TB patients. It will explore the factors of success of TB treatment using inter-disciplinary approach, integrating social sciences and economic analyses into TB research. The project is composed of 3 comprehensive phases:

* Phase 1: baseline assessment of the TB situation.
* Phase 2: anthropological study, investigating various domains contributing to patients cure using a range of qualitative research methods. At the end of this investigation, it is expected that determinants of care will be clearly identified. On this basis, suitable methods for improving patients' adherence to treatment will be tailored and developed.
* Phase 3: these methods will be tested and compared using a cluster randomised controlled trial design, in populations served by defined health centres. Their efficacy will be measured in terms of improvement of the classical TB control programme indicators (cure rate, defaulter rate, failure rate, death rates). The methods will also be evaluated on their acceptability by the TB patients and the communities and on their feasibility (duration : 24 months).

Expected results:

Methods to improve patients' adherence to treatment that are affordable, acceptable and sustainable will be developed and tested according to qualitative and quantitative criteria.

DETAILED DESCRIPTION:
General Project Methods

The proposed research seeks to develop and test innovative methods to improve treatment success rates in TB patients in Senegal. It will explore the factors of success of TB treatment using inter-disciplinary approach, integrating social sciences and economic analyses into TB research. The project is composed of 3 comprehensive phases, that will be run concurrently and complement each other:

* Phase 1: baseline assessment of the TB situation. It is first proposed to assess the magnitude of the TB problem and of the means to control it through a standard baseline assessment (6 months).
* Phase 2: anthropological study, investigating various domains contributing to patients cure (the patients, the community, the general health services, the policy makers and the TB control staff), using a range of qualitative research methods (12 months). At the end of this investigation, it is expected that determinants of care will be clearly identified with a comprehensive understanding of their relation/interface. On this basis, suitable methods for improving patients' adherence to treatment will be developed.
* Phase 3: these methods will be tested and compared using a cluster randomised controlled trial design, in populations served by defined health centres. Their efficacy will be measured in terms of improvement of the classical TB control programme indicators (cure rate, defaulter rate, failure rate, death rates). The methods will also be evaluated on their acceptability by the TB patients and the communities and on their feasibility (24 months).

Methods of the Intervention Trial:

The intervention is intended to improve access to care and increase adherence to treatment, targeting simultaneously DHC staff, TB patients and communities, and includes four components:

1. improving communication between health personnel and patients through appropriate training;
2. decentralising treatment to remote health posts and involving community health workers (CHW);
3. strengthening the DOT strategy by giving patients the opportunity to choose their treatment supporter; and
4. reinforcing supervision of health posts by the DHC team.

The intervention is applied at the District Health Centre (DHC) level, which is the unit of randomisation.

Sample Size:

Based on the detection of an average of 100 new TB cases per DHC per year, an estimated coefficient of variability k=0.12, an estimated success rate in the control arm of 65% using conventional TB control programmes procedures, with 80% power and a type I error of 5%, the required sample size aiming to detect a difference of at least 15% in the treatment success rate between the intervention and control arms is eight DHCs per arm. In order to take into account the variation in recruitment of TB patients between the DHCs, the randomisation is stratified on baseline detection rate of sputum smear positive cases in 2001, that were classified as less than 60/100 000 and more than or equal to 60/100 000.

Patients and follow-up DHCs with a functional TB diagnosis and treatment unit, where no other research projects were being undertaken, were eligible for inclusion. The study population consisted of all individuals presenting to the DHC between June 2003 and May 2004 with newly diagnosed sputum-smear positive pulmonary TB (at least two positive specimens), aged 15 years or more, and living in the district served by the DHC. Written informed consent was obtained at recruitment and patients were followed-up during the course of their eight month treatment regimen, with the last patients seen in January 2005.

Smear-negative and extra-pulmonary tuberculosis cases, as well as re-treatment cases, were not eligible for the study. Patients were recruited into the study between June 2003 and May 2004 and followed up till January 2005.

Endpoints:

Primary endpoints are both the proportion of recruited patients experiencing treatment success (those cured + those completing treatment), and the proportion of patients defaulting from treatment before completion. A "cured" patient is defined by a negative sputum-smear at eight months and on at least one previous occasion. Patients "completing treatment" are those missing smear results but who had finished their treatment regimen. A "defaulter" is defined as a patient who definitely stopped treatment before completion.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed sputum-smear positive pulmonary TB (at least two positive specimens), aged 15 years or more, and living in the district served by the District Health Centre.

Exclusion Criteria:

* Smear-negative tuberculosis cases
* extra-pulmonary tuberculosis cases
* TB re-treatment cases

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2003-05; Study Completion 2005-01

PRIMARY OUTCOMES:
TB treatment success rate (cure + completed treatment)
Treatment defaulting rates

SECONDARY OUTCOMES:
treatment failure rate
death rate

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha Ndir, MD, Principal Investigator — Programme de Lutte anti-tuberculeuse, Dakar, Senegal; Christian Lienhardt, MD, Principal Investigator — Institut de Recherche pour le Developpement, Paris, France
Locations (1):
- Programme National de Lutte Anti-tuberculeuse, Dakar, Senegal

REFERENCES:
- [Background] Lienhardt C, Ogden JA. Tuberculosis control in resource-poor countries: have we reached the limits of the universal paradigm? Trop Med Int Health. 2004 Jul;9(7):833-41. doi: 10.1111/j.1365-3156.2004.01273.x. PMID 15228495
- [Derived] Thiam S, LeFevre AM, Hane F, Ndiaye A, Ba F, Fielding KL, Ndir M, Lienhardt C. Effectiveness of a strategy to improve adherence to tuberculosis treatment in a resource-poor setting: a cluster randomized controlled trial. JAMA. 2007 Jan 24;297(4):380-6. doi: 10.1001/jama.297.4.380. PMID 17244834